CLINICAL TRIAL: NCT00738530
Title: A Randomised, Double-blind Study to Evaluate the Efficacy and Safety of Avastin Plus Roferon Compared With Placebo Plus Roferon on Overall Survival and Tumor Assessment in Nephrectomised Patients With Metastatic Clear Cell Renal Cell Carcinoma
Brief Title: A Study of Avastin (Bevacizumab) Added to Interferon Alfa-2a (Roferon) Therapy in Patients With Metastatic Renal Cell Cancer With Nephrectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BO17705; 2004-000282-35 (EudraCT Number)
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Results first posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-05

CONDITIONS: Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Bevacizumab; Interferon alpha-2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Bevacizumab + IFN-Alfa-2A (Experimental): Bevacizumab infusions will be administered every 2 weeks at a dose of 10 milligram per kilogram (mg/kg) for 52 weeks or until disease progression or unacceptable toxicity. Interferon alfa-2a (IFN-Alfa-2A) will be administered 3 times per week as a subcutaneous injection at a dose of 9 million international units (MIU) for 52 weeks or until disease progression or major toxicity.
  Interventions: Drug: Bevacizumab [Avastin]; Drug: Interferon alfa 2a [Roferon]
- Placebo + IFN-Alfa-2A (Placebo Comparator): Placebo matched with Bevacizumab infusions will be administered every 2 weeks for 52 weeks or until disease progression or unacceptable toxicity. IFN-Alfa-2A will be administered 3 times per week as a subcutaneous injection at a dose of 9 MIU for 52 weeks or until disease progression or major toxicity.
  Interventions: Drug: Interferon alfa 2a [Roferon]; Drug: Placebo

INTERVENTIONS:
Drug: Bevacizumab [Avastin] — 10 mg/kg IV every 2 weeks
  Arms: Bevacizumab + IFN-Alfa-2A
Drug: Interferon alfa 2a [Roferon] — 9 MIU SC 3 times/week
Drug: Placebo — IV every 2 weeks
  Arms: Placebo + IFN-Alfa-2A

SUMMARY:
This 2-arm study will evaluate the efficacy and safety of Avastin versus placebo in combination with Roferon as first-line treatment in participants with metastatic renal cell cancer (clear cell type) who have had nephrectomy. The anticipated time of study treatment is 1-2 years, and the target sample size is greater than (>)500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* metastatic renal cell cancer (clear cell type);
* nephrectomy;
* absence of proteinuria.

Exclusion Criteria:

* prior systemic treatment for metastatic renal cell cancer;
* major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to study treatment start;
* presence of brain metastases or spinal cord compression;
* ongoing need for full dose anticoagulants;
* uncontrolled hypertension;
* clinically significant cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 649 (Actual)
Dates: Start 2004-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (89):
- Australia (8):
  - Adelaide
  - Brisbane
  - Canberra
  - Frankston
  - Kurralta Park
  - Melbourne
  - Perth
  - Sydney
- Belgium (3):
  - Antwerp
  - Brussels
  - Wilrijk
- Czechia (4):
  - Chomutov
  - České Budějovice
  - Hradec Králové
  - Pilsen
- Finland (2):
  - Tampere
  - Turku
- France (16):
  - Angers
  - Bordeaux
  - Caen
  - Clermont-Ferrand
  - Grenoble
  - Lille
  - Limoges
  - Lyon
  - Marseille
  - Nice
  - Poitiers
  - Saint-Herblain
  - Strasbourg
  - Suresnes
  - Toulouse
  - Villejuif
- Germany (8):
  - Berlin
  - Darmstadt
  - Hamburg
  - Hanover
  - Mannheim
  - Marburg
  - München
  - Planegg
- Hungary (2):
  - Budapest
  - Szombathely
- Israel (5):
  - Holon
  - Ramat Gan
  - Rehovot
  - Tel Aviv
  - Ẕerifin
- Italy (8):
  - Livorno
  - Milan
  - Modena
  - Napoli
  - Perugia
  - Roma
  - Rozzano
  - Torino
- Netherlands (2):
  - Amsterdam
  - Nijmegen
- Norway (4):
  - Ålesund
  - Oslo
  - Stavanger
  - Trondheim
- Poland (6):
  - Bydgoszcz
  - Krakow
  - Lodz
  - Olsztyn
  - Tarnów
  - Warsaw
- Russia (3):
  - Moscow
  - Obninsk
  - Saint Petersburg
- Singapore, Singapore
- Spain (8):
  - Barcelona
  - Granada
  - Madrid
  - Málaga
  - Pontevedra
  - Santander
  - Valencia
  - Zaragoza
- Switzerland (3):
  - Basel
  - Bern
  - Geneva
- Taiwan (4):
  - Chang Gung
  - Kaohsiung City
  - Taichung
  - Taipei
- United Kingdom (2):
  - London
  - Manchester

REFERENCES:
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 821 participants were screened for this study, and 649 of these were randomized to receive double-blind treatment.
Groups:
- Bevacizumab + IFN-Alfa-2A: Bevacizumab infusions were administered every 2 weeks at a dose of 10 milligram per kilogram (mg/kg) for 52 weeks or until disease progression or unacceptable toxicity. Interferon alfa-2a (IFN-Alfa-2A) was administered 3 times per week as a subcutaneous injection at a dose of 9 million international units (MIU) for 52 weeks or until disease progression or major toxicity.
- Placebo + IFN-Alfa-2A: Placebo matched with Bevacizumab infusions were administered every 2 weeks for 52 weeks or until disease progression or unacceptable toxicity. IFN-Alfa-2A was administered 3 times per week as a subcutaneous injection at a dose of 9 MIU for 52 weeks or until disease progression or major toxicity.
Period: Overall Study
Arm/Group | Bevacizumab + IFN-Alfa-2A | Placebo + IFN-Alfa-2A
Started | 327 | 322
Treated | 325 | 316
Completed | 93 | 84
Not Completed | 234 | 238
Not completed — Death | 220 | 224
Not completed — Lost to Follow-up | 8 | 6
Not completed — Withdrawal by Subject | 6 | 8

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population (ITT) included all participants randomized into the study.
Groups:
- Bevacizumab + IFN-Alfa-2A: Bevacizumab infusions were administered every two weeks at a dose of 10 mg/kg for 52 weeks or until disease progression or unacceptable toxicity. IFN-Alfa-2A was administered 3 times per week as a subcutaneous injection at a dose of 9 MIU for 52 weeks or until disease progression or major toxicity.
- Placebo + IFN-Alfa-2A: Placebo matched with Bevacizumab infusions were administered every two weeks for 52 weeks or until disease progression or unacceptable toxicity. IFN-Alfa-2A was administered 3 times per week as a subcutaneous injection at a dose of 9 MIU for 52 weeks or until disease progression or major toxicity.
- Total: Total of all reporting groups
Arm/Group | Bevacizumab + IFN-Alfa-2A | Placebo + IFN-Alfa-2A | Total
Number analyzed (Participants) | 327 | 322 | 649
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (10.12) | 59.4 (10.89) | 59.7 (10.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 87 | 192
  Male | 222 | 235 | 457

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Died
Time Frame: Baseline up to 4.25 years
Population: ITT population included all participants randomized into the study.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + IFN-Alfa-2A | Placebo + IFN-Alfa-2A
Number analyzed (Participants) | 327 | 322
percentage of participants | 67.3 | 69.6

2. Primary Outcome: Overall Survival (OS) Duration
Description: Duration of survival was defined as the time between the date of randomization and date of death due to any cause. Participants still alive at the time of analysis were censored at the date they were last known to be alive. Kaplan-Meier estimates were used for analysis.
Time Frame: Baseline until death (up to 4.25 years)
Population: ITT population included all participants randomized into the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + IFN-Alfa-2A | Placebo + IFN-Alfa-2A
Number analyzed (Participants) | 327 | 322
months | 23.3 [20.4 to 27.0] | 21.3 [18.4 to 24.5]
Statistical Analysis 1: Comparison: Bevacizumab + IFN-Alfa-2A vs Placebo + IFN-Alfa-2A; Test type: Superiority or Other; p = 0.3360, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.76 to 1.10]

3. Secondary Outcome: Percentage of Participants With Disease Progression or Death
Description: Progressive disease was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the appearance of one or more new lesions and/or the unequivocal progression of existing non-target lesions.
Time Frame: Baseline until disease progression or death, whichever occurred first (assessed at baseline, Weeks 8, 16, 24, 32, 44, 56, 68 thereafter every 12 weeks up to week 104 and then every 6 months up to 4.25 years)
Population: ITT population included all participants randomized into the study.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + IFN-Alfa-2A | Placebo + IFN-Alfa-2A
Number analyzed (Participants) | 327 | 322
percentage of participants | 92.0 | 92.5

4. Secondary Outcome: Progression Free Survival (PFS) According to Modified Response Evaluation Criteria in Solid Tumors (mRECIST)
Description: Progression-free survival was defined as the time between the date of randomization and the first date of documented progression or date of death due to any cause, whichever occurred first. Tumor assessment was performed using modified RECIST. Progressive disease was defined as at least a 20 percentage(%) increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the appearance of one or more new lesions and/or the unequivocal progression of existing non-target lesions. Participants without an event were censored at the date of last follow-up for progression or date of last available tumor measurement if no follow-up assessment for progression was performed. Participants who were randomized but not exposed to study drug and had no further follow-up were censored on the day of randomization.
Time Frame: as for outcome 3
Population: ITT population included all participants randomized into the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + IFN-Alfa-2A | Placebo + IFN-Alfa-2A
Number analyzed (Participants) | 327 | 322
months | 10.2 [7.7 to 11.1] | 5.5 [4.2 to 5.7]
Statistical Analysis 1: Comparison: Bevacizumab + IFN-Alfa-2A vs Placebo + IFN-Alfa-2A; Test type: Superiority or Other; p = 0.0004, Log Rank; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.64 to 0.88]

5. Secondary Outcome: Time to Progression (TTP) According to Modified Response Evaluation Criteria in Solid Tumors (mRECIST)
Description: Time to progression was defined as the time between date of randomization and date of documented progression. Tumor assessment was performed using mRECIST. Progressive disease was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the appearance of one or more new lesions and/or the unequivocal progression of existing non-target lesions. Participants without an event (including participants who died before progressive disease) were censored at the date of last follow-up for progression or date of last available tumor measurement if no follow-up assessment for progression was performed. Participants who were randomized but not exposed to study drug and had no further follow-up were censored on the day of randomization.
Time Frame: as for outcome 3
Population: ITT population included all participants randomized into the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + IFN-Alfa-2A | Placebo + IFN-Alfa-2A
Number analyzed (Participants) | 327 | 322
months | 10.2 [7.9 to 11.6] | 5.5 [4.3 to 5.8]
Statistical Analysis 1: Comparison: Bevacizumab + IFN-Alfa-2A vs Placebo + IFN-Alfa-2A; Test type: Superiority or Other; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.62 to 0.86]

6. Secondary Outcome: Percentage of Participants With Treatment Failure
Description: Treatment failure is defined as insufficient therapeutic response (including disease progression), death, withdrawal of treatment due to adverse events or laboratory abnormality, or withdrawal of informed consent. Tumor assessment was performed using mRECIST. Progressive disease was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the appearance of one or more new lesions and/or the unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 3
Population: ITT population included all participants randomized into the study.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + IFN-Alfa-2A | Placebo + IFN-Alfa-2A
Number analyzed (Participants) | 327 | 322
percentage of participants | 90.5 | 91.6

7. Secondary Outcome: Time to Treatment Failure (TTF) According to Modified Response Evaluation Criteria in Solid Tumors (mRECIST)
Description: Time to treatment failure was defined as the time between the date of randomization and the date of insufficient therapeutic response (including disease progression), death, withdrawal of treatment due to adverse events or laboratory abnormality, or withdrawal of informed consent. Tumor assessment was performed using mRECIST. Progressive disease was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the appearance of one or more new lesions and/or the unequivocal progression of existing non-target lesions. Participants without an event were censored at the date of last tumor assessment or last treatment administration, whichever occurred last. Participants who were randomized but not exposed to study drug and had no further follow-up were censored on the day of randomization.
Time Frame: as for outcome 3
Population: ITT population included all participants randomized into the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + IFN-Alfa-2A | Placebo + IFN-Alfa-2A
Number analyzed (Participants) | 327 | 322
months | 8.1 [7.1 to 10.2] | 4.5 [3.8 to 5.6]
Statistical Analysis 1: Comparison: Bevacizumab + IFN-Alfa-2A vs Placebo + IFN-Alfa-2A; Test type: Superiority or Other; p = 0.0023, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.66 to 0.92]

8. Secondary Outcome: Percentage of Participants With Objective Response According to mRECIST
Description: Objective response referred to participants with complete response (CR) or partial response (PR). CR: disappearance of all target lesions, non-target lesions, and normalization of tumor marker level. PR: greater than or equal to (>=) 30% decrease in sum of the longest diameter (LD) of all target lesions taking as reference the screening sum LD. To be assigned a status of PR or CR, changes in tumor measurements had to be confirmed by repeat assessments that should have been performed no less than 4 weeks after the criteria for response were first met. Longer intervals as determined by the study protocol were also appropriate.
Time Frame: as for outcome 3
Population: ITT population included all participants randomized into the study. Number of participants analyzed (N) = participants with measurable disease at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + IFN-Alfa-2A | Placebo + IFN-Alfa-2A
Number analyzed (Participants) | 306 | 289
percentage of participants | 32.4 | 12.5
Statistical Analysis 1: Comparison: Bevacizumab + IFN-Alfa-2A vs Placebo + IFN-Alfa-2A; Test type: Superiority or Other; p < .0001, Chi-squared; Difference in response rates = 19.90, 95% CI 2-sided [13.2 to 26.6]

9. Secondary Outcome: Percentage of Participants With Best Overall Response According to Modified Response Evaluation Criteria in Solid Tumors (mRECIST)
Description: Best response recorded from the start of treatment until disease progression. Based on assessment of CR, PR, stable disease (SD), or progressive disease (PD), according to mRECIST. CR: disappearance of all target lesions, non-target lesions, and normalization of tumor marker level. PR: >=30% decrease under baseline of the sum of the LD of all target lesions. CR and PR persist on repeat imaging study at least 4 weeks after initial documentation. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Reference is the smallest sum LD. PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the appearance of one or more new lesions and/or the unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 3
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + IFN-Alfa-2A | Placebo + IFN-Alfa-2A
Number analyzed (Participants) | 306 | 289
percentage of participants
  Complete Response (CR) | 1.6 | 2.4
  Partial Response (PR) | 30.7 | 10.0
  Stable Disease (SD) | 44.4 | 50.5
  Progressive Disease (PD) | 20.6 | 33.2
  Missing (no response assessment) | 2.6 | 3.8

10. Secondary Outcome: Change From Baseline in Karnofsky Performance Status
Description: Karnofsky performance score is used to quantify participant's general well-being and activities of daily life and participants were classified based on their functional impairment. Karnofsky performance score is 11 level score which ranges between 0 (death) to 100 (no evidence of disease). Higher score means higher ability to perform daily tasks.
Time Frame: Baseline, Week 7, 15, 23, 31, 43
Population: Safety population: all participants randomized and exposed to study drug (8 randomized participants did not receive study treatment and were not included, 2 in bevacizumab and 6 in placebo group). 12 participants randomized to placebo received bevacizumab, were included in bevacizumab arm. n=number of evaluable participants at specified time point.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Bevacizumab + IFN-Alfa-2A | Placebo + IFN-Alfa-2A
Number analyzed (Participants) | 337 | 304
score on a scale
  Baseline (n=337, 304) | 90 [70 to 100] | 90 [70 to 100]
  Change at Week 7 (n=291, 263) | 0 [-50 to 10] | 0 [-60 to 20]
  Change at Week 15 (n=242, 196) | 0 [-40 to 20] | 0 [-60 to 20]
  Change at Week 23 (n=195, 143) | 0 [-90 to 20] | 0 [-60 to 20]
  Change at Week 31 (n=166, 108) | 0 [-40 to 20] | 0 [-50 to 20]
  Change at Week 43 (n=137, 79) | 0 [-40 to 20] | 0 [-20 to 10]

ADVERSE EVENTS:
Time Frame: Baseline up to 4.25 years
Description: Safety population: all participants randomized and exposed to study drug (8 randomized participants did not receive study treatment and were not included, 2 in bevacizumab and 6 in placebo group). 12 participants randomized to placebo received bevacizumab, were included in bevacizumab arm. n=number of evaluable participants at specified time point.
Arm/Group | Bevacizumab + IFN-Alfa-2A | Placebo + IFN-Alfa-2A
Serious Adverse Events (participants affected / at risk) | 103/337 | 51/304
Other Adverse Events (participants affected / at risk) | 319/337 | 279/304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + IFN-Alfa-2A (N=337) | Placebo + IFN-Alfa-2A (N=304)
Pneumonia (Infections and infestations) | 8 | 0
Gastroenteritis (Infections and infestations) | 3 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Infection anal abscess (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 0
Postoperative abscess (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 0
Renal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 7 | 0
Pyrexia (General disorders) | 5 | 0
Asthenia (General disorders) | 2 | 2
General physical health (General disorders) | 2 | 0
Deterioration pain (General disorders) | 0 | 2
Adverse drug reaction (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Injection site reaction (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Necrosis (General disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Epilepsy (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Gliosis (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Hyperaesthesia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Leukoencephalopathy (Nervous system disorders) | 1 | 0
Movement disorder (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 3
Depression (Psychiatric disorders) | 4 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Mood altered (Psychiatric disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 0
Hypotension (Vascular disorders) | 0 | 2
Aneurysm ruptured (Vascular disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pyrophosphate muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephritic syndrome (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Benign penile neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Medical device complication (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Postoperative wound (Injury, poisoning and procedural complications) | 1 | 0
Complication traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Skin graft failure (Skin and subcutaneous tissue disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Hypercalcaemia of malignancy (Endocrine disorders) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Retinal vein thrombosis (Eye disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + IFN-Alfa-2A (N=337) | Placebo + IFN-Alfa-2A (N=304)
Pyrexia (General disorders) | 149 | 130
Asthenia (General disorders) | 108 | 83
Fatigue (General disorders) | 107 | 83
Influenza like illness (General disorders) | 84 | 78
Chills (General disorders) | 53 | 54
Mucosal inflammation (General disorders) | 18 | 11
Nausea (Gastrointestinal disorders) | 97 | 78
Diarrhoea (Gastrointestinal disorders) | 70 | 48
Vomiting (Gastrointestinal disorders) | 47 | 42
Constipation (Gastrointestinal disorders) | 39 | 25
Abdominal pain (Gastrointestinal disorders) | 28 | 25
Abdominal pain upper (Gastrointestinal disorders) | 23 | 13
Stomatitis (Gastrointestinal disorders) | 17 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 63 | 41
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 | 28
Back pain (Musculoskeletal and connective tissue disorders) | 38 | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 | 21
Bone pain (Musculoskeletal and connective tissue disorders) | 23 | 15
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 25 | 13
Anorexia (Metabolism and nutrition disorders) | 122 | 93
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 90 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 45 | 38
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 39
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 17 | 0
Headache (Nervous system disorders) | 82 | 50
Dizziness (Nervous system disorders) | 27 | 27
Dysgeusia (Nervous system disorders) | 21 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 32 | 23
Pruritus (Skin and subcutaneous tissue disorders) | 30 | 20
Alopecia (Skin and subcutaneous tissue disorders) | 24 | 19
Rash (Skin and subcutaneous tissue disorders) | 17 | 21
Anaemia (Blood and lymphatic system disorders) | 33 | 39
Neutropenia (Blood and lymphatic system disorders) | 23 | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 21 | 13
Hypertension (Vascular disorders) | 95 | 27
Depression (Psychiatric disorders) | 38 | 30
Insomnia (Psychiatric disorders) | 21 | 20
Anxiety (Psychiatric disorders) | 9 | 18
Weight decreased (Investigations) | 68 | 44
Proteinuria (Renal and urinary disorders) | 68 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.